CLINICAL TRIAL: NCT07100821
Title: Thoracic Fluid Content as an Outcome Predictor in Respiratory Intensive Care Unit
Brief Title: Thoracic Fluid Content as an Outcome Predictor in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer faculty of medicine, Mansoura University Hospital
Other Study IDs: MS.19.12.354
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Diseases
Keywords: Thoracic fluid content; respiratory intensive care unit
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients indicated for admission to respiratory critical care unit of chest medicine department: 130 patients >18 years old were enrolled during the period from December 2023 to December 2024
  Interventions: Diagnostic Test: Hemodynamic parameters was measured by using electric cardiometry (ICON)

INTERVENTIONS:
Diagnostic Test: Hemodynamic parameters was measured by using electric cardiometry (ICON) — Hemodynamic parameters was measured daily at 10 a.m by using ICON non-invasive cardiometer model C3 made in Germany by OSYPKA medical (figure 5) by placing the four sensors on the neck and left side of the thorax allow for the continuous measurement of the changes of electrical conductivity within the thorax parameters such as CO, TFC, SVV and FTC were calculated 3 times with 5-min intervals and stored on the device automatically.

SUMMARY:
Hemodynamic monitoring is measuring and monitoring the factors that influence the force and flow of the blood. It is an important aspect of patients care in operating rooms and critical care units. It aims to guide medical management so as to prevent or treat organ failure and improve the outcomes of patients.

DETAILED DESCRIPTION:
Hemodynamic monitoring is measuring and monitoring the factors that influence the force and flow of the blood. It is an important aspect of patients care in operating rooms and critical care units. It aims to guide medical management so as to prevent or treat organ failure and improve the outcomes of patients. This monitoring itself includes several different techniques and may range from invasive to less and even non-invasive techniques.

Critically ill patients are often hemodynamically unstable (or at risk of becoming unstable) owing to hypervolemia, cardiac dysfunction or alterations of vasomotor function, leading to organ dysfunction, deterioration into multi-organ failure and eventually death range from 15% to 25% of patients admitted to intensive care units.

Impedance cardiography (ICG) and Electrical Cardiometry (EC) are recently developed technologies to measure thoracic fluid content (TFC), cardiac output (CO) and other hemodynamic parameters. Both ICG and EC derive CO from measurements of Thoracic Electrical Bioimpedance (TEB).

One of the parameters examined by electrical cardiometry is thoracic fluid content(TFC) ,which is inversely associated with the patient's transthoracic electrical bioimpedance, and reflects the total (intravascular and extravascular) fluid volume contained in the chest cavity. A study concluded that electrical cardiometry monitoring indicated new possibility to anticipate prognosis of pneumonia patient. Increased thoracic fluid content value would relate to worse outcome of the patient like mortality and intensive care unit admission. Electrical cardiometry monitoring allows real-time measurements of thoracic fluid content without restraining the patient or invasive catheters.

In ARDS patients with cardiac comorbidities, TFC can distinguish between non-cardiogenic and cardiogenic pulmonary edema. In addition, TFC is helpful in the differential diagnosis of the mechanisms of respiratory failure. Thus, recently it was shown that TFC was greater in ARDS than in patients with atelectasis or pleural effusion. Therefore, depending on the TFC value, we can provide different therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Patients indicated for admission to respiratory critical care unit of chest medicine department at Mansoura University Hospitals whatever the indication was.

Exclusion Criteria:

* Patients with malignancy either primary or metastatic lung cancer.
* Advanced chronic pulmonary fibrosis.
* Pleural and or pericardial effusions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any Patient indicated for admission to respiratory critical care unit of chest medicine department at Mansoura University Hospitals whatever the indication was
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
length of respiratory intensive care unit stay | 6 months
  Thoracic fluid content as an outcome predictor in length of stay in respiratory intensive care unit
duration of invasive mechanical ventilation | 6 months
  Thoracic fluid content as an outcome predictor in duration of invasive mechanical ventilation

SECONDARY OUTCOMES:
mortality | 12 months
  Thoracic fluid content and hemodynamic parameters measurement as an outcome predictor in mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No